CLINICAL TRIAL: NCT00165581
Title: A Pilot Clinical Trial to Evaluate High Dose Rate Intracavitary Brachytherapy as the Sole Method of Radiation Therapy for Favorable Stage I and II Breast Cancer
Brief Title: High Dose Rate Intracavitary Brachytherapy as the Sole Method of Radiation Therapy for Breast Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to continuing review
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-259
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Breast Cancer
Keywords: Intracavitary brachytherapy; radiation therapy; Stage I breast cancer; Stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Brachytherapy

INTERVENTIONS:
Device: High Dose Intracavitary Brachytherapy

SUMMARY:
The purpose of this study is to understand the side effects (skin reaction, infection and abscess formation) at the site of radiation treatment, which my occur during the treatment and following 2 months using a new method of radiation therapy for breast cancer.

DETAILED DESCRIPTION:
* Radiation treatment will be delivered in an outpatient setting, twice a day in 5 consecutive treatment days. There will be a minimum 6-hour interval between the two daily treatments. The applicator is a simple tube with an inflatable balloon at one end, a channel in the middle of the tube for treatment, and two adapters at the other end.
* Following surgical removal of the breast cancer, the radiation oncologist with the assistance of the surgeon or radiologist will place the applicator in the surgical cavity. A small radioactive source, iridium-192, will be inserted into the applicator by a special machine and after the final treatment, the applicator will be removed.
* The following procedures will be done while the patient is on radiation therapy: post-partial mastectomy mammogram of micro-calcifications to confirm complete removal; CT scans for radiation treatment planning; monitoring of the skin for side effects; photographs of the breasts prior to the surgery, prior to placement of the applicator and at 60 days after radiation treatment to evaluate the cosmetic outcome of the treatment.
* Participation in this study will last approximately 2 months after completion of radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* AJCC stage I or II histologically confirmed invasive ductal carcinoma of the breast with a lesion < or = to 3cm, treated with partial mastectomy
* 45 years of age or older
* Negative inked pathologic specimen
* > or = to 3mm margins of partial mastectomy or re-excision specimen to be confirmed prior to introducing radiation source
* Negative post-partial mastectomy or post re-excision mammography if cancer presented with malignancy-associated microcalcifications; no remaining suspicious microcalcifications in the breast before brachytherapy
* Invasive ductal, medullary, papillary, colloid, or tubular histologies
* Time interval from final definitive breast surgical procedure to brachytherapy treatment is less than 8 weeks

Exclusion Criteria:

* Distant metastases
* Invasive lobular carcinoma or pure ductal carcinoma in situ or nonepithelial breast malignancies such as sarcoma or lymphoma
* Proven multifocal, multicentric carcinoma with other clinically or radiologically suspicious areas in the ipsilateral breast unless confirmed to be negative for malignancy by biopsy
* Pregnant or lactating
* Confirmed positive axillary nodes in the ipsilateral axilla. Palpable or radiographically suspicious contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes, unless there is histologic confirmation that these nodes are negative for tumor
* Prior non-hormonal therapy for the present breast cancer, including radiation therapy and chemotherapy
* Collagen vascular diseases, specifically systemic lupus erythematosis, scleroderma, keloid, ataxia, telangiectasia, or dermatomyositis
* Co-existing medical condition in whom life expectancy is < 2 years
* Psychiatric or addictive disorders
* Paget's disease of the nipple
* Skin involvement regardless of size
* Breast unsatisfactory for brachytherapy
* Surgical margins which cannot be microscopically assessed or are positive at pathological evaluation
* Extensive intraductal carcinoma
* Any previously treated contralateral breast carcinoma or synchronous bilateral breast carcinoma
* Other malignancy, except non-melanoma skin cancer, < 5 years prior to participation in this study
* Diffuse suspicious microcalcifications

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2002-12; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the technical feasibility and acute 60-day toxicity of intracavitary HDR brachytherapy when used as the sole method of radiation therapy for patients with Stage I and II breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip M. Devlin, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts